CLINICAL TRIAL: NCT07064850
Title: Vasomotor Symptoms in Post-Hysterectomy Women With Ovarian Conservation: A Prospective Study
Brief Title: Vasomotor Symptoms in Post-Hysterectomy Women With Ovarian Conservation
Status: Enrolling by invitation | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Professor, Northwestern University
Other Study IDs: STU00223626
Record Dates: First submitted 2025-07-07; First posted 2025-07-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Vasomotor Symptoms
Keywords: Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to learn about vasomotor symptoms (such as hot flashes and night sweats) in the short-term period after a hysterectomy.

The main question it aims to answer is: How common and severe are vasomotor symptoms shortly after surgery in people who have had a hysterectomy?

Participants will complete a survey before surgery to assess baseline symptoms, and again 2 weeks after surgery to see if there are any changes.

DETAILED DESCRIPTION:
Hysterectomies are among the most common surgical procedures for women in the United States, with approximately 600,000 operations performed annually. Traditionally, it has been assumed that retaining one or both ovaries during hysterectomy mitigates the onset and severity of vasomotor symptoms, such as hot flashes and night sweats. However, recent research indicates that even with ovarian conservation, women may experience a higher incidence of persistent vasomotor symptoms compared to those who have not had the surgery. These symptoms can significantly impact quality of life, underscoring the need for comprehensive studies that track the progression of vasomotor symptoms post-hysterectomy. Despite their clinical importance, the precise timeline of symptom onset and the influence of ovarian retention remain poorly understood.

Existing studies on surgical menopause primarily focus on factors such as depression, anxiety, and abdominal pain. No study to date has followed women from the immediate postoperative period through the subsequent months to assess the onset, type, and frequency of vasomotor symptoms. Additionally, research on surgical menopause often lacks detailed information on the diagnostic indications for hysterectomy and fails to differentiate between women who retained both ovaries versus those who retained only one at the time of surgery. This study aims to provide a better understanding of the relationship between the onset and severity of vasomotor symptoms in order to improve postoperative care, guide patient counseling, and develop targeted interventions to mitigate vasomotor symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. 35-50 years old
2. Undergoing hysterectomy with at least one ovary conserved
3. Ability to provide informed consent

Exclusion Criteria:

(None specified)

Ages: 35 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — cisgender women
Study Population: The study population will consist of patients scheduled for hysterectomy with ovarian conservation at an urban academic medical center. Participants will be recruited from the surgical gynecology service.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Changes in Vasomotor Symptom Frequency | Baseline period to 2 weeks pre-operative
  One primary outcome measure is the change in average vasomotor symptom frequency score from baseline (pre-operative) to 2 weeks post-operative. The symptoms evaluated will be hot flashes, night sweats, increased sweating, sleep disturbances, and heart palpitations. Participants will rate how often they experience each symptom: never, rarely, sometimes, or often. For each symptom, average scores at baseline will be compared to scores collected 2 weeks after surgery to assess changes in symptom frequency.
Changes in Vasomotor Symptom Distress | Baseline period to 2 weeks pre-operative
  One primary outcome measure is the change in average vasomotor symptom distress scores from baseline (pre-operative) to 2 weeks post-operative. The symptoms assessed will include hot flashes, night sweats, increased sweating, sleep disturbances, and heart palpitations. Participants will rate how bothersome each symptom is using a 7-point Likert scale (0 = not at all bothersome, 6 = extremely bothersome). For each symptom, average distress scores at baseline will be compared to those collected 2 weeks post-operatively to evaluate changes in perceived symptom burden. Higher scores indicate greater symptom distress.

SECONDARY OUTCOMES:
Thematic Analysis of Patient-Reported Symptom Experiences | Baseline period to 2 weeks post-operative
  This secondary outcome measure involves the qualitative analysis of patient comments related to symptom experiences. Participants will have the option to provide open-ended feedback in both the pre-operative and post-operative surveys. The qualitative data will focus on the same vasomotor symptoms assessed quantitatively (hot flashes, night sweats, increased sweating, sleep disturbances, and heart palpitations), as well as any additional symptoms reported after surgery. Patient narratives will be analyzed using thematic analysis to identify recurring themes and the overall impact of symptoms on daily life. This qualitative component is intended to provide contextual depth to the quantitative symptom distress scores.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy P Milad, MD MS, Principal Investigator — Northwestern Medicine
Locations (1):
- Northwestern University, Chicago, Illinois, United States